CLINICAL TRIAL: NCT01240720
Title: A Phase I/II Dose Finding and Efficacy Study of the Tumour Targeting Human 131I-F16SIP Monoclonal Antibody in Patients With Cancer
Brief Title: A Dose Finding and Efficacy Study of the Tumour Targeting Human 131I-F16SIP Monoclonal Antibody in Patients With Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: Eudax S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-F16SIPI131-06/07
Record Dates: First submitted 2010-10-27; First posted 2010-11-15 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Cancer
Keywords: I131; F16; antibody; monoclonal; tumor targeting; radioimmunotherapy; lymphoma, breast and lung cancer; Patients with different cancer types
MeSH Terms: conditions — Neoplasms; Lymphoma; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I131-F16SIP (Experimental): Phase I: Multicentre, open-label, two-step singlearm dose escalation study in sequential cohorts of patients with cancer.
  Phase II: Prospective, open-label, single-arm, multicentre study of 131I-F16SIP, given at the RD of 55.5 mCi/m2, as determined in phase I.
  Interventions: Drug: 131I-F16SIP Radioimmunotherapy (RIT)

INTERVENTIONS:
Drug: 131I-F16SIP Radioimmunotherapy (RIT) — * Dosimetric evaluation with 131I-F16SIP or 124I-F16SIP will be performed to assess eligibility for Radioimmunotherapy.
  * Patients eligible for Radioimmunotherapy will receive 55.5 mCi/m2 as established in the Phase I part of the study. A single dose of 5 to 10 mg of 131I-F16SIP will be administered intravenously (I.V).

SUMMARY:
The aim of this Study Protocol is to provide a basis for the clinical development of 131I-F16SIP as an anti-cancer therapeutic agent.

The study follows and is greatly motivated by the promising results of a Phase I/II study with a similar investigational drug developed by our Company, 131I-L19SIP, in several Italian centers.

DETAILED DESCRIPTION:
The F16SIP antibody is a fully human antibody, capable of preferential localization around tumour blood vessels while sparing normal tissues. The formation of new blood vessels is a rare event in the adult (exception made for the female reproductive cycle), but is a pathological feature of most aggressive types of cancer. The study aims at determining the therapeutic potential of the F16 antibody in SIP format,labelled with the radionuclide 131I, for the treatment of patients with different cancer types.

ELIGIBILITY:
Inclusion Criteria:

1. Phase I:

   Patients with cancer, with progressive disease in pre-study period, refractory to conventional standard treatments.

   Solid Tumor: Histologically/cytologically confirmed diagnosis of cancer, preferably lung cancer, prostate cancer or colorectal cancer (CRC). At least one measurable (minimum 2.0 cm), non irradiated lesion defined according to modified RECIST criteria i.e. whenever the measurable disease is restricted to a solitary lesion, its neoplastic nature need not be confirmed by cytology/histology.

   Lymphoproliferative Diseases: Histologically/cytologically confirmed diagnosis of lymphoproliferative disease. At least one measurable (minimum 2.0 cm) non irradiated lesion defined according to modified RECIST criteria, i.e. whenever the measurable disease is restricted to a solitary lesion; its neoplastic nature needs to be confirmed by cytology/histology.

   Phase II:

   Patients with lymphoma, breast cancer or lung cancer with progressive disease in pre-study period, refractory to conventional standard treatments, will be enrolled in the study. Presence of brain metastases at time of screening does not represent an exclusion criterion. Lesions will be evaluated according to RECIST for solid tumors or to the Revised response criteria for malignant lymphoma (Cheson BD, JCO 2007, 25, 579-58) for lymphomas.
2. ECOG performance status grade 0 or 1.
3. Age ≥18.
4. Adequate haematological, liver and renal function (haemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1.50 x 109/L; platelets ≥ 100 x 109/L, bilirubin within UNL; alkaline phosphatase≤ 2.5 x UNL; ALT, AST ≤ UNL or ≤ 2.5 x UNL in case of liver metastases; albumin ≥ 2.5 g/dL; creatinine ≤ UNL.
5. All acute toxic effects (excluding alopecia) of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v.3.0) Grade ≤ 1.
6. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment.
7. If of childbearing potential, agreement to use adequate contraceptive methods (e.g., oral contraceptives, condoms, or other adequate barrier controls, intrauterine contraceptive devices, or sterilization) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
8. Evidence of a personally signed and dated IEC-approved Informed Consent indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the study.
9. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.
10. Life expectancy of at least 3 months.
11. Signed and dated informed consent.

Exclusion Criteria:

1. Chemotherapy, radiation, hormonotherapy or immunotherapy or participation in any investigational drug study within 4 weeks of RIT treatment at the RD (6 weeks in case of prior nitroureas chemotherapy).
2. Prior radiation dose > 30% of bone marrow volume.
3. Presence of cirrhosis or active hepatitis.
4. Presence of serious cardiac (congestive heart failure, heart insufficiency > grade II NYHA, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorders.
5. Presence of uncontrolled intercurrent illness or any condition which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study.
6. Recovery from major trauma including surgery within 4 weeks of administration of study treatment.
7. Pregnancy or lactation or unwillingness to use adequate method of birth control.
8. Active infection or incomplete wound healing.
9. Known history of allergy to intravenously administered proteins / peptides / antibodies.
10. Any conditions that in the opinion of the investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-09; Primary Completion 2011-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum tolerated Dose | 4 weeks
  Establishment of the maximum tolerated dose (MTD), a recommended dose (RD) for the phase II part, and the safety of dosimetric and therapeutic administration of escalating dosages of the human radiolabeled antibody 131I-F16SIP.
Phase II: Antitumour activity | 14 months
  Investigation of the antitumour activity of 131I-F16SIP at the RD.

SECONDARY OUTCOMES:
Phase I: Study of the variation of radioactivity of 131I or 124I in whole blood, at several time intervals (Pharmacokinetics) | 2 days
  Evaluation of the pharmacokinetics of 131I-F16SIP and 124I-F16SIP.
Phase II: Adverse Events as a Measure of Safety | 30 days/ administration
  Determination of the overall safety profile of the iodinated antibody characterized by type, frequency, severity, timing and relationship to study therapy of adverse events and laboratory abnormalities in the first and eventual following administrations in all patients receiving a therapeutic dose.
Phase II: Overall Response Rate (ORR) | 6 and 12 months
  Evaluation of the overall Response Rate (ORR) for all patients having received a therapeutic dose.
Phase II: Progression free survival (PFS) | 6 and 12 months
  Evaluation of the progression free survival (PFS) for all patients having received a therapeutic dose.
Phase II: Survival rate | 6 and 12 months
  Evaluation of the survival rate at 6 and 12 months and overall survival time for all patients having received a therapeutic dose.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, Dr, Principal Investigator — IRST (Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori)
Locations (6):
- Italy (6):
  - University Hospital Pisa, Pisa, Tuscany
  - Policlinico S. Orsola-Malpighi- Azienda Ospedaliero-Universitaria di Bologna, Bologna
  - ASUR Zona Territoriale 9, Medicina Nucleare Ospedale di Macerata, Macerata
  - Irst - Istituto Scientifico Romagnolo Per Lo Studio E La Cura Dei Tumori - Meldola (Fc), Meldola
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale Di Napoli, Napoli
  - Arcispedale Santa Maria Nuova Di Reggio Emilia, Reggio Emilia